CLINICAL TRIAL: NCT04692311
Title: Motivation, Usability and Functionality of an Intelligent Activity-based Client-centred Training System in Neurological Rehabilitation: a Pilot Study
Brief Title: Pilot Study Concerning an Intelligent Activity-based Client-centred Training System in Neurorehabilitation
Acronym: i-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PXL University College (Other)
Collaborators: Hasselt University (Other); Hogeschool West-Vlaanderen (Unknown); Jessa Hospital (Other); Ziekenhuis Oost-Limburg (Other); Revalidatie & MS Centrum Overpelt (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Els Knippenberg, Researcher, PXL University College
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: i-ACT pilot
Record Dates: First submitted 2020-12-21; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Central Nervous System Diseases; Neurological Rehabilitation
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Mixed-method pilot study in which persons with central nervous system diseases and occupational therapists were included
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persons with central nervous system diseases (Experimental): Persons with central nervous system diseases received additional training with i-ACT during 6 weeks. After final training, a semi-structured interview was performed. And at six weeks follow-up, a final assessment took place.
  Interventions: Device: an intelligent client-centred task-oriented training; Other: Semi-structured interview
- Occupational therapists (Other): Occupational therapists were invited to a semi-structured interview to gather information about their professional opinion regarding i-ACT.
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Device: an intelligent client-centred task-oriented training — 3 x 45min of training with i-ACT system
  Other Names: i-ACT
  Arms: Persons with central nervous system diseases
Other: Semi-structured interview — Participants, patients and therapists, were invited to a semi-structured interview after training period.

SUMMARY:
The pilot study was performed to evaluate the usability, credibility and expectancy of an intelligent, activity-based client-centred training system (i-ACT), and the motivation towards its use in neurological rehabilitation over a short period of time.

DETAILED DESCRIPTION:
A mixed-method study was performed in four rehabilitation centres in Belgium. An homogenous convenience sample was recruited among persons with central nervous system disorders.

Participants received 3 x 45 minutes of training with the i-ACT system during six weeks, additional to conventional care. The Canadian Occupational Performance Measure (COPM) was used to collect and evaluate patients' individual goals towards rehabilitation. These goals were discussed with the therapists before implementing movements and exercises for each patient in the i-ACT system.

The following demographic data were obtained from the medical files: age, gender, and diagnosis. Outcomes measures were collected at baseline (T0), after 2 (T1), 4 (T2) and 6 (T3) weeks of training and at 9 weeks follow-up (T4).

The primary outcome measures were the Intrinsic Motivation Inventory (IMI), the System Usability Scale (SUS), Credibility/Expectancy Questionnaire (CEQ), the Canadian Occupational Performance Measure (COPM), and Wolf Motor Function Test (WMFT). The secondary measures were the Manual Ability Measure-36 (MAM-36), Modified Fatigue Impact Scale (MFIS), Trunk Impairment Scale (TIS), and Active Range of Motion (AROM).

After final training with i-ACT, a semi-structured interview was performed to gather more information about the participants' perception towards i-ACT.

For quantitative data, within-group differences of all the assessments were analysed using Friedman's ANOVA and Wilcoxon signed-rank test. Alpha was set at 0.05; No Bonferroni correction was applied as it is not compulsory in an exploratory study and furthermore, results are regarded as hypothesis for further investigations.

The qualitative data was collected and recorded with a voice recorder. No specific analysis was used as the interview collected data to support or oppose the findings of the quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* a medical diagnosis of central nervous system disease
* dysfunction in upper limb and/or core stability
* Persons with multiple sclerosis (MS) had to be free of treatment with corticosteroids for one month.
* Persons with stroke or spinal cord injury, had to be at least three months post injury.

Exclusion Criteria:

* severe spasticity (when spasticity impedes movement)
* severe cognitive impairment (person is not able to understand and follow instructions)
* severe communicative impairment (person is not able to answer questions)
* severe visual impairment (person is not able to see the television screen)
* persons who use an electric wheelchair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Intrinsic Motivation Inventory | 2 weeks
  Motivation towards a therapy, in this i-ACT
Intrinsic Motivation Inventory | 4 weeks
  Motivation towards a therapy, in this i-ACT
Intrinsic Motivation Inventory | 6 weeks
  Motivation towards a therapy, in this i-ACT
Intrinsic Motivation Inventory | 12 weeks (i.e. 6 weeks follow-up)
  Motivation towards a therapy, in this i-ACT
System Usability Scale | 2 weeks
  Usability of a system, in this i-ACT. Range of scores from 0 (negative) to 100 (positive).
System Usability Scale | 4 weeks
  Usability of a system, in this i-ACT. Range of scores from 0 (negative) to 100 (positive).
System Usability Scale | 6 weeks
  Usability of a system, in this i-ACT. Range of scores from 0 (negative) to 100 (positive).
System Usability Scale | 12 weeks (i.e. 6 weeks follow-up)
  Usability of a system, in this i-ACT. Range of scores from 0 (negative) to 100 (positive).
Credibility/Expectancy Questionnaire | 2 weeks
  Credibility and expectancy of a training system, in this i-ACT. The range of scores on each subscale (i.e. credibility and expectancy) is 27.
Credibility/Expectancy Questionnaire | 4 weeks
  Credibility and expectancy of a training system, in this i-ACT. The range of scores on each subscale (i.e. credibility and expectancy) is 27.
Credibility/Expectancy Questionnaire | 6 weeks
  Credibility and expectancy of a training system, in this i-ACT. The range of scores on each subscale (i.e. credibility and expectancy) is 27.
Credibility/Expectancy Questionnaire | 12 weeks (i.e. 6 weeks follow-up)
  Credibility and expectancy of a training system, in this i-ACT. The range of scores on each subscale (i.e. credibility and expectancy) is 27.
Canadian Occupational Performance Measure | Baseline
  By means of a semi-structured interview, participants are asked to identify their 5 main goals in self-care, productivity and/or leisure.
  Scores range from 0 to 10 (best score) in each defined goal.
Canadian Occupational Performance Measure | 4 weeks
  By means of a semi-structured interview, participants are asked to identify their 5 main goals in self-care, productivity and/or leisure.
  Scores range from 0 to 10 (best score) in each defined goal.
Canadian Occupational Performance Measure | 6 weeks
  By means of a semi-structured interview, participants are asked to identify their 5 main goals in self-care, productivity and/or leisure.
  Scores range from 0 to 10 (best score) in each defined goal.
Canadian Occupational Performance Measure | 12 weeks (i.e. 6 weeks follow-up)
  By means of a semi-structured interview, participants are asked to identify their 5 main goals in self-care, productivity and/or leisure.
  Scores range from 0 to 10 (best score) in each defined goal.
Wolf Motor Function Test | Baseline
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).
Wolf Motor Function Test | 2 weeks
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).
Wolf Motor Function Test | 4 weeks
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).
Wolf Motor Function Test | 6 weeks
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).
Wolf Motor Function Test | 12 weeks (i.e. 6 weeks follow-up)
  Arm-hand functioning. The test contains 17 items and are scored from 0 (not able to perform tesk) to 5 (normal performance).

SECONDARY OUTCOMES:
Manual Ability Measure-36 | Baseline
  Manual ability. Scores range from 0 (impossible to perform) to 4 (easy to perform)
Manual Ability Measure-36 | 2 weeks
  Manual ability. Scores range from 0 (impossible to perform) to 4 (easy to perform)
Manual Ability Measure-36 | 4 Weeks
  Manual ability. Scores range from 0 (impossible to perform) to 4 (easy to perform)
Manual Ability Measure-36 | 6 weeks
  Manual ability. Scores range from 0 (impossible to perform) to 4 (easy to perform)
Manual Ability Measure-36 | 12 weeks (i.e. 6 weeks follow-up)
  Manual ability. Scores range from 0 (impossible to perform) to 4 (easy to perform)
Modified Fatigue Impact Scale | Baseline
  Fatigue. Twenty-one items ar scored on a 5-point Likert scale (range from 0, never, to 4, almost always). The higher the score the most impact fatigue has on the life of the person. .
Modified Fatigue Impact Scale | 2 weeks
  Fatigue. Twenty-one items ar scored on a 5-point Likert scale (range from 0, never, to 4, almost always). The higher the score the most impact fatigue has on the life of the person. .
Modified Fatigue Impact Scale | 4 weeks
  Fatigue. Twenty-one items ar scored on a 5-point Likert scale (range from 0, never, to 4, almost always). The higher the score the most impact fatigue has on the life of the person. .
Modified Fatigue Impact Scale | 6 weeks
  Fatigue. Twenty-one items ar scored on a 5-point Likert scale (range from 0, never, to 4, almost always). The higher the score the most impact fatigue has on the life of the person. .
Modified Fatigue Impact Scale | 12 weeks (i.e. 6 weeks follow-up)
  Fatigue. Twenty-one items ar scored on a 5-point Likert scale (range from 0, never, to 4, almost always). The higher the score the most impact fatigue has on the life of the person. .
Trunk Impairment Scale | Baseline
  Trunk impairment. Scores range from 0 (minimum) to 23. The higher the score the less motor impairment is present in the trunk.
Trunk Impairment Scale | 2 weeks
  Trunk impairment. Scores range from 0 (minimum) to 23. The higher the score the less motor impairment is present in the trunk.
Trunk Impairment Scale | 4 weeks
  Trunk impairment. Scores range from 0 (minimum) to 23. The higher the score the less motor impairment is present in the trunk.
Trunk Impairment Scale | 6 weeks
  Trunk impairment. Scores range from 0 (minimum) to 23. The higher the score the less motor impairment is present in the trunk.
Trunk Impairment Scale | 12 weeks (i.e. 6 weeks follow-up)
  Trunk impairment. Scores range from 0 (minimum) to 23. The higher the score the less motor impairment is present in the trunk.
Active Range of Motion | Baseline
  Active range of motion
Active Range of Motion | 2 weeks
  Active range of motion
Active Range of Motion | 4 weeks
  Active range of motion
Active Range of Motion | 6 weeks
  Active range of motion
Active Range of Motion | 12 weeks (i.e. 6 weeks follow-up)
  Active range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Spooren, Prof.Dr, Study Chair — PXL University College

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request, the data (in Dutch) can be shared with other researchers.